CLINICAL TRIAL: NCT04635982
Title: Kinesiotape on Quadriceps and Gluteus in Counter Movement Jump and Sprint in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina Abellan, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48490314N
Record Dates: First submitted 2020-11-11; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Sports Physical Therapy; Athletics; Performance
Keywords: Kinesiotape; Soccer; Sprint

STUDY DESIGN:
Intervention Model Description: Thirty-seven subjects were randomly allocated to the different study groups using the software AleatorMetod.xls. Subjects were divided into three groups: 13 subjects were assigned to the experimental group with KT activation (KTact); 12 subjects, to the placebo group with a sham tape KT (KTst); and 12 subjects, to the control group (CG).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): With regard to the Kinesiotape technique, 2 I-shaped tapes were placed at the quadriceps, following the same direction of the muscle fibres and with no tension. At the gluteus, 2 I-shaped tapes were applied following the same direction of the muscle fibres and with no tension.
  Interventions: Other: Kinesiotape of the physical performance
- Experimental Group (Experimental): In rectus femoris, origin was under the anterosuperior iliac spines, and taping finished with a Y-shape pattern under the patella. After that, an I-shaped KT was applied over vastus medialis and vastus lateralis muscles in both quadriceps. Finally, subjects were taped with a Y-shaped KT at the gluteus maximus muscles. Tape tension was between 25% and 50%.
  Interventions: Other: Kinesiotape of the physical performance
- Control Group (No Intervention): It has not done any intervention in this group.

INTERVENTIONS:
Other: Kinesiotape of the physical performance — It has done a countermovement vertical jump, a twenty meter sprint and a kinesio tape application technique
  Arms: Experimental Group; Placebo Group

SUMMARY:
The main objective of this study is to analyse the effect of KT on countermovement jump (CMJ) and sprint immediately and 24 hours after its application on the quadriceps and gluteus maximus.

DETAILED DESCRIPTION:
Kinesiotape (KT) is a technique commonly used in sports practice. It may be beneficial in enhancing muscle function by additional cutaneous afferent stimulation. The objective of this study was to analyze the effect of KT on countermovement jump (CMJ) and 20-m sprints immediately and 24 hours after its application on the quadriceps and gluteus maximus. A total of 37 male soccer players (19.7 ± 0.9 years old) were randomly assigned to one of 3 groups: experimental group: KT activation (KTact), placebo group: sham tape (KTst), and control group (CG). Participants performed a 30-minute preliminary warm-up, after which they conducted CMJ and 20-m sprint tests. These tests were repeated later (with KT application or not) and after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* soccer players;
* age of 18-25 years;
* a regular attendance at training sessions

Exclusion Criteria:

* history of L1-L5 radiculopathy or lumbo-sacral pathology ;
* any treatment with KT on quadriceps or gluteus in the month prior to the study;
* history of systemic diseases that may affect the nervous system, musculoskeletal injuries or surgeries in the lower limb during the year prior to the study;
* use of analgesics or nonsteroidal anti-inflammatory drugs.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Countermovement vertical jump | 24 hours
  Countermovement jump test was carried out on a Chronojump Boscosystem® contact platform and the jump height was measured in centimeters
20 m sprints test | 24 hours
  Sprint-speed measurements were conducted using Chronojump

CONTACTS AND LOCATIONS:
Overall Officials: Javier Reina Abellan, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Maria Cinta Gomez, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The timing of the application of KT in the gluteus maximus and the quadriceps should be taken into account as the speed of execution in football players decreases immediately after its application and 24 hours after the test is performed